CLINICAL TRIAL: NCT04297293
Title: Effects of Ramosetron Orally Disintegrating Tablet on the Prophylaxis of Postdischarge Nausea and Vomiting in High-risk Patients Undergoing Day Surgery Under General Anesthesia
Brief Title: Ramosetron OD Tablet and Postdischarge Nausea and Vomiting
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Jung Shin, Associate Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B-2002/594-003
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Day Surgery
MeSH Terms: interventions — ramosetron

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ramosetron-ODT (Experimental)
  Interventions: Drug: Ramosetron
- Control (No Intervention)

INTERVENTIONS:
Drug: Ramosetron — Ramosetron orally disintegrating tablet 0.1 mg is administered after discharge (postoperative day 1 and day 2)
  Arms: Ramosetron-ODT

SUMMARY:
Postoperative nausea and vomiting after general anesthesia is one of the common anesthetic complications. If the patient is discharged from the hospital after surgery, proper treatment may be delayed or impossible if nausea and vomiting occurred. Thus, it is necessary to prevent these symptoms beforehand. Patients who underwent day-surgery will be treated with prophylactic ramosetron orally disintegrating tablets to determine whether the frequency of nausea and vomiting is decreased when the patient returned home after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo day-surgery under general anesthesia and are discharged on the day of surgery

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patients who are taking other serotonin receptor antagonists
* Patients who have galactose intolerance or Lapp lactase deficiency
* patients who have glucose-galactose malabsorption

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
The change in the occurrence of postoperative nausea | Postoperative 30 minute, 3 hour, 24 hour, and 48 hour
The change in the occurrence of postoperative vomiting | Postoperative 30 minute, 3 hour, 24 hour, and 48 hour

SECONDARY OUTCOMES:
The change in the severity of postoperative nausea | Postoperative 30 minute, 3 hour, 24 hour, and 48 hour
  Numerical rating scale range from 0 to 100 (0 = no pain, 100 = the most severe pain imaginable)
The change of patient's satisfaction score | Postoperative 30 minute, 3 hour, 24 hour, and 48 hour
  Numerical rating scale range from 0 to 100 (0 = no pain, 100 = the most severe pain imaginable)
The change in the number of postoperative administration of rescue antiemetic drug | Postoperative 30 minute, 3 hour, 24 hour, and 48 hour

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Jung Shin, MD., PhD., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

REFERENCES:
- [Derived] Shin HJ, Park YH, Chang M, Chae YJ, Lee HT, Lee OH, Min SK, Do SH. Effects of ramosetron orally disintegrating tablets on the prophylaxis of post-discharge nausea and/or vomiting in female patients undergoing day surgery under general anesthesia: a randomized controlled trial. Perioper Med (Lond). 2022 May 12;11(1):17. doi: 10.1186/s13741-022-00251-6. PMID 35546414